CLINICAL TRIAL: NCT02194478
Title: Pilot Study of a Brief Mind/Body Meditation Intervention for Allina Health Employees
Brief Title: Stress Reduction for Busy Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S091301
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Stress
Keywords: Stress; Meditation; Mind body
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 8 Week Meditation (Other): Allina Health employees undergoing 8 week meditation intervention
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — 30 minute, 8 week meditation

SUMMARY:
This is a pre-post intervention pilot study to evaluate the impact of a 30-minute, 8-week mind-body/meditation intervention on self-reported quality of life in individuals employed by Allina Health. Outcomes will include validated questionnaires for depressive symptomology, perceived stress, anxiety, healthy lifestyle, quality of life as well as biological outcomes of salivary cortisol for a sub-sample of employees.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years
* Actively-working healthcare professional employed by Allina Health.

Exclusion Criteria:

* Previous participation in an Allina Health stress reduction program
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Perceived stress change from baseline at week 8 | Baseline, Week 8
  Perceived stress will be measured through the Perceived Stress Scale at baseline and week 8.

SECONDARY OUTCOMES:
Salivary Cortisol Levels Change from baseline at week 8 | Baseline, Week 8
  Salivary samples will be obtained at baseline and week 8.
Lifestyle Profile change from baseline at week 8 | Baseline, Week 8
  The Lifestyle Profile questionnaire measures self actualization, health responsibility, exercise, nutrition, interpersonal support, and stress management. It will be administered at baseline and week 8.
Work productivity and activity impairment change from baseline at week 8 | Baseline, Week 8
  Work productivity and activity impairment will be measured through the WPAI:GH and will be administered at baseline and week 8.
Promis-29 score change from baseline at week 8 | Baseline, Week 8
  The Promis-29 is a 29 item questionnaire measuring physical function, fatigue, pain, depression, anxiety, and social role participation. The questionnaire will be administered at baseline and week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Dusek, PhD, Principal Investigator — Allina Health
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States